CLINICAL TRIAL: NCT07036068
Title: A Clinical Study on the Use of a Domestically Produced Cryoablation System Combined With Balloon Cryoablation Technology for the Treatment of Paroxysmal Atrial Fibrillation
Acronym: Balloon cryoab
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort EP MedTech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Gao Henggan, Cui Kaijun, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: West China Hospital（Sichuan）
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Paroxysmal Atrial Fibrillation (PAF)
Keywords: PFA; PeAF; PFA/RF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-centre, post-marketing study (Experimental): This study aims to evaluate the safety and efficacy of using a domestically produced cardiac cryoablation system to treat paroxysmal atrial fibrillation.
  Interventions: Device: IceMagic™ CryoAblation Catheter

INTERVENTIONS:
Device: IceMagic™ CryoAblation Catheter — IceMagic™ CryoAblation Catheter is available in two diameters: 23 mm and 28 mm. Each diameter has two types of balloon outer surfaces: with or without multi-channel tissue temperature measurement function. The catheter length is 140 cm, and the tube diameter is 10.5 F. Doctors can choose according to the size of the target pulmonary vein.

SUMMARY:
To validate the safety and efficacy of balloon cryoablation technology and the accompanying disposable intracardiac mapping electrode catheter and adjustable guide sheath for the treatment of paroxysmal atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age between 18 and 80 years old, male or non-pregnant female.
2. Confirmed diagnosis of paroxysmal atrial fibrillation requiring cryoablation surgery.
3. Fully understands the treatment plan and voluntarily signs the informed consent form, willing to undergo the examinations, surgery, and follow-up required by the plan.

Exclusion Criteria:

1. Patients who have undergone atrial fibrillation ablation surgery
2. Reproductive-age patients who cannot use effective contraception within 12 months of enrolment
3. Left atrial size ≥50 mm, left ventricular ejection fraction ≤40%
4. Left atrial thrombus
5. Patients who have undergone atrial septal defect repair surgery or atrial myxoma
6. Patients with cerebrovascular disease within the past 3 months (including stroke or transient ischaemic attack)
7. Patients with cardiovascular events within the past 3 months (including acute myocardial infarction, coronary artery intervention or bypass surgery, artificial valve replacement or repair, or atrial or ventricular incision)
8. Patients with acute or severe systemic infection
9. Patients with severe liver or kidney disease
10. Patients with a significant tendency to bleed or haematological disorders
11. Patients with malignant tumours or end-stage diseases
12. Patients deemed ineligible for this trial by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Three-month follow-up success rate after surgery | Three months after surgery
  Postoperative 3-month treatment success rate: Specifically refers to the proportion of participants who, during the 3-month follow-up period post-surgery (after the washout period), did not experience any episodes of atrial fibrillation/atrial flutter/atrial tachycardia lasting ≥30 seconds, as confirmed by electrocardiogram (ECG), Holter monitoring, or equivalent rhythm monitoring methods (including single-lead ECG), without the use of Class I or Class III antiarrhythmic drugs, relative to the total number of enrolled participants.

SECONDARY OUTCOMES:
Immediate ablation success rate | On the 1 day of the surgery
  This refers to the proportion of subjects who achieved electrical isolation after surgery among the total number of patients enrolled in the study. The verification method involves waiting for 20 minutes after successful pulmonary vein electrical isolation and then reconfirming pulmonary vein conduction block.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China